CLINICAL TRIAL: NCT03387358
Title: Nasal Bridle Assessment in the Intensive Care Unit: An Observational Study to Examine the Effectiveness and Adverse Events of the Nasal Bridle Securement Device in High Risk ICU Patients
Brief Title: An Observational Study Examining Adverse Events and Effectiveness of the Nasal Bridle Securement Device in ICU Patients
Acronym: NBA-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Providence Healthcare (Other)
Responsible Party: Principal Investigator, Vininder K. Bains, Principal Investigator, University of British Columbia
Other Study IDs: H16-03176
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Enteral Nutrition
Keywords: intensive care unit; nasal bridle securement device; small bore feeding tube; adverse events; enteral nutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Historical Comparison Group: This group includes patients who were admitted to St. Paul's Hospital ICU (Vancouver BC, Canada) from September 2014 to September 2015, and had a small bore feeding tube in place at some point during their ICU admission, and were matched to key variables to the prospective observational treated group.
- Prospective Observational Treated Group: This group includes all patients who were admitted to St. Paul's Hospital ICU from Nov. 2017 to Dec. 2018, and nasal bridle securement device for small bore feeding tubes at some point during their ICU admission. The clinical indicators for a nasal bridle securement device outlined in our nursing practice standards include one or more of the following: recurrent nasoenteric tube dislodgement; confused and/or agitated patients; fluoroscopically or endoscopically placed nasoenteric tube; history of difficult tube placement; facial burn victims with nasoenteric tube; and/or oily skin causing decreased adhesion of traditional securement.
  Interventions: Device: Nasal bridle securement device for small bore feeding tubes

INTERVENTIONS:
Device: Nasal bridle securement device for small bore feeding tubes — A Nasal bridle securement device is an alternative method to securing small bore feeding tubes which are most commonly secured with adhesive tape to the nose. A nasal bridle securement device instead secures the feeding tube to a cloth ribbon that is inserted in one nostril, over then nasal bridle and out the other nostril.
  Other Names: AMTBridle TM: Nasal Tube Retaining System
  Groups: Prospective Observational Treated Group

SUMMARY:
Nasal bridle securement device (NBSD) is a device used to keep feeding tubes in place. Unlike tape, it keeps tubes in place by tying the feeding tube to a fabric string that is looped in through one nostril, over the nasal bridge and out the other nostril. The purpose of this study is to measure how effective a NBSD is at keeping feeding tubes in place and what effect that will have on how many calories ICU patients receive. Also, the another objective is to measure what, if any, harmful or undesirable outcomes happen with using a NBSD in our ICU patients.

DETAILED DESCRIPTION:
BACKGROUND/JUSTIFICATION: Adequate nutritional support is an important part of treatment in critical illness. It is usually delivered via a nasoenteric feeding tube because ICU patients may have an altered level of consciousness, delirium, and/or dependence on mechanical ventilation. Feeding tubes are traditionally secured with adhesive tape, making dislodgement of the tube possible. Dislodgement of feeding tubes can lead to suboptimal caloric intake and increased risk of aspiration of feeds/pneumonia. An alternative to this is the nasal bridle securement device (NBSD), which has been shown to have lower rates of tube dislodgement, but the evidence is limited as it is a relatively new medical device. There is also little documented about any adverse events associated with use of the NBSD.

Prior to 2016, all small bore feeding tubes inserted in ICU patients at St. Paul's Hospital were secured with adhesive tape exclusively. The ICU team began using NBSD in 2016 only in patients who were at higher risk for, or with, tube dislodgement. The clinical indications outlined in our Nursing Practice Standards (i.e., "Nursing Practice Standard NCS5652 - Nasal Bridle") are: recurrent nasoenteric tube dislodgement, confused and/or agitated patients, fluoroscopically or endoscopically placed nasoenteric tube, history of difficult tube placement, facial burn victims with nasoenteric tube and/or oily skin causing decreased adhesion of traditional securement.

PURPOSE: The purpose of this study is three-fold, in patients who demonstrated a higher risk for, or with, tube dislodgement: to describe the incidence and characteristics of adverse events associated with NBSD; to examine the effectiveness of the NBSD at prevention of inadvertent dislodgement; to assess if use of this devise is associated with a difference in the proportion of total caloric goal delivered.

RESEARCH QUESTIONS:

1. To determine the incidence and characteristics of all types of adverse events associated with the use of NBSD to secure small bore feeding tubes in ICU patients who have demonstrated a high risk for, or with, tube dislodgement.
2. To determine if there is a difference in the rate of inadvertent dislodgement of small bore feeding tubes in ICU patients who demonstrate a high risk for, or with, tube dislodgement between ICU patients whose feeding tube is secured with a NBSD versus those who were secured with tape. Rate of tube dislodgement is defined as number of tube dislodgements per total number ICU days with a small bore feeding tube in place.

   Null hypothesis: there is no difference in the rate of inadvertent tube dislodgement.

   Alternate hypothesis: there is a difference in the rate of inadvertent tube dislodgement.
3. To determine if there is a difference in the proportion of total caloric goals delivered in ICU patients with small bore feeding tubes with a high risk for or with tube dislodgement in ICU patients whose feeding tube is secured with a NBSD versus those who were secured with tape.

Null hypothesis: there is no difference in the proportion of total caloric goals delivered.

Alternate hypothesis: there is a difference in the proportion of total caloric goals delivered.

RESEARCH DESIGN: The prospective observational treated group will include all ICU patients who required a NBSD securement for their feeding tube as per standard practice (i.e., PHC Nursing Practice Standard NCS5652 - Nasal Bridle) from when ethics and operational approvals are obtained until December 31, 2018.

A historical comparison group will be selected from patients admitted to ICU between September 1, 2014 and September 30, 2015 (prior to use of NBSD in the ICU) who have a small bore feeding tube and match key variables.

Since the NBSD is used only in a selected number of ICU patients, in order to select an equivalent sample for the historical comparison group, the investigators will use the ICU database to identify key variables for matching. The patients who were admitted to the ICU from October 1, 2016 until October 30, 2017 and had a small bore feeding tube will be the Interim Group. Using the ICU Database, a statistical comparison of variables in patients from the Interim Group who had, versus did not have, a NBSD to secure their small bore feeding tube will be used to identify what key variables should be used for selecting the historical comparison group.

INCLUSION/EXCLUSION CRITERIA: Inclusion criteria for both the historical and prospective groups are: Admitted to the ICU at St. Paul's Hospital; had a small bore feeding tube in place during their ICU admission.

In addition, the prospective observational treated group will also need to have a NBSD inserted at some time during their ICU admission as per the criteria outlined in the Nursing Practice Standard NCS5652. These clinical indicators include: recurrent nasoenteric tube dislodgement, confused and/or agitated patients, fluoroscopically or endoscopically placed nasoenteric tube, history of difficult tube placement, facial burn victims with nasoenteric tube and/or oily skin causing decreased adhesion of traditional securement. The historical comparison group only need to have a small bore feeding tube, secured by tape, and are matched by key variables.

For both the prospective observational treated group and the historical comparison group who were admitted to the ICU and had a small bore feeding tube in place during their ICU admission, the only patients who are excluded are:

1. those where were not permitted to be fed by the gastrointestinal system (as per Doctor's Orders);
2. and/or did not meet the criteria for use of a NBSD as per the "Nursing Practice Standard NCS5652 - Nasal Bridles"

MEASUREMENT: Demographic data (i.e., age, gender, comorbidities etc.), diagnosis and admission history (i.e., admission date, diagnoses, length of stay, feeding tube placement etc.) will be used to describe and compare the historical comparison group and the prospective observational treated group. To address the first research question regarding adverse events, all types of adverse events associated with the use of the NBSD will be recorded, including adverse events associated with its insertion, use, and removal. To address the second research question regarding inadvertent dislodgement, both the number of inadvertent dislodgements, and duration of tube retainment will be compared between the treated and historical comparison group. To address the third research question regarding caloric intake, the proportion of daily total caloric goal delivered will be compared between the treated and historical comparison group.

DATA COLLECTION: There are three sources of data for this study. The ICU Database has data from every admitted ICU patient. It includes demographic data, diagnoses, admission history, information on a number of procedures and interventions like the use of small bore feeding tubes, patient assessments, and patient outcomes. The ICU Nasal Bridle Database collects information for every ICU patient which has a NBSD inserted (see "Nasal Bridle Tracker Form" attached in Section 9.8.B.). It records data on insertion details, removal details and additional information on adverse event or other issues. The patient chart will be reviewed to collect additional information about the caloric goals and actual total caloric intake. See the NBA-ICU Data Collection Form (Section 9.8.A.) for further details.

STATISTICAL ANALYSIS: Descriptive statistics will be used to compare demographic variables between the prospective observational treated group and the historical comparison group. All types of adverse events including unintentional tube dislodgement, events associated with insertion, use or removal of the NBSD and all other will be qualitatively and quantitatively described. The Goodness of Fit Test or the non-parametric equivalent (Fisher's Exact Test) will be used to assess if there is a difference in the rate of inadvertent dislodgement. The Student T Test will be used to assess if there is a difference in proportion of total caloric goal delivered between treated and historical comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for both the historical and prospective groups are: Admitted to the ICU at St. Paul's Hospital; had a small bore feeding tube in place during their ICU admission.

In addition, the prospective observational treated group will also need to have a NBSD inserted at some time during their ICU admission as per the criteria outlined in the Nursing Practice Standard NCS5652. These clinical indicators include: recurrent nasoenteric tube dislodgement, confused and/or agitated patients, fluoroscopically or endoscopically placed nasoenteric tube, history of difficult tube placement, facial burn victims with nasoenteric tube and/or oily skin causing decreased adhesion of traditional securement.

The historical comparison group only need to have a small bore feeding tube, secured by tape, and are matched by key variables.

Exclusion Criteria:

* For both the prospective observational treated group and the historical comparison group who were admitted to the ICU and had a small bore feeding tube in place during their ICU admission, the only patients who are excluded are:

  1. those where were not permitted to be fed by the gastrointestinal system (as per Doctor's Orders);
  2. and/or did not meet the criteria for use of a NBSD as per the Nursing Practice Standard NCS5652

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the ICU at St. Paul's Hospital in Vancouver BC between September 1 2014 and September 30, 2015 OR October 1, 2017 and December 31, 2018 and had a small bore feeding tube in place as a standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2019-02-24 (Estimated); Study Completion 2019-02-24 (Estimated)

PRIMARY OUTCOMES:
Incidence and characteristics of all types of adverse events | During the ICU admission (up to 4 weeks)
  Describe the prevalence and characteristics of all types of adverse events associated with use of the Nasal Bridle Securement device, including with its insertion, use and removal.

SECONDARY OUTCOMES:
Rate of inadvertent dislodgement of a small bore feeding tube while in the ICU | During the ICU admission (up to 4 weeks)
  the rate of inadvertent dislodgement is defined as the number of inadvertent tube per total ICU days with a small bore feeding tube (i.e., number of dislodgment/ICU days with small bore feeding tube)
Proportion of total daily caloric goal delivered. | Measured daily for the duration of the ICU admission (up to 4 weeks)
  This is the proportion of total daily caloric goal that was actually received by the participant (i.e., 100 x actual caloric intake/goal caloric intake). Calories are measured in kilocalories (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Aeberhardt, RD, Principal Investigator — Providence Healthcare
Locations (1):
- Providence Health Care, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beavan J, Conroy SP, Harwood R, Gladman JR, Leonardi-Bee J, Sach T, Bowling T, Sunman W, Gaynor C. Does looped nasogastric tube feeding improve nutritional delivery for patients with dysphagia after acute stroke? A randomised controlled trial. Age Ageing. 2010 Sep;39(5):624-30. doi: 10.1093/ageing/afq088. Epub 2010 Jul 27. PMID 20667840
- [Background] Bechtold ML, Nguyen DL, Palmer LB, Kiraly LN, Martindale RG, McClave SA. Nasal bridles for securing nasoenteric tubes: a meta-analysis. Nutr Clin Pract. 2014 Oct;29(5):667-71. doi: 10.1177/0884533614536737. PMID 25606648
- [Background] Brandt CP, Mittendorf EA. Endoscopic placement of nasojejunal feeding tubes in ICU patients. Surg Endosc. 1999 Dec;13(12):1211-4. doi: 10.1007/pl00009623. PMID 10594268
- [Background] Brugnolli A, Ambrosi E, Canzan F, Saiani L; Naso-gastric Tube Group. Securing of naso-gastric tubes in adult patients: a review. Int J Nurs Stud. 2014 Jun;51(6):943-50. doi: 10.1016/j.ijnurstu.2013.12.002. Epub 2013 Dec 25. PMID 24440003
- [Background] Nasal Bridle Devices for the Securement of Nasoenteric Feeding Tubes in Adult Patients: Comparative Clinical Effectiveness, Safety, and Cost-Effectiveness [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2016 Dec 19. Available from http://www.ncbi.nlm.nih.gov/books/NBK424238/ PMID 28211665
- [Background] Jackson RS, Sharma S. Retained nasal tube bridle system insertion stylet presenting as nasal foreign body: a report of two cases. Am J Otolaryngol. 2015 Mar-Apr;36(2):296-8. doi: 10.1016/j.amjoto.2014.10.033. Epub 2014 Nov 5. PMID 25465320
- [Background] Lamont T, Beaumont C, Fayaz A, Healey F, Huehns T, Law R, Lecko C, Panesar S, Surkitt-Parr M, Stroud M, Warner B. Checking placement of nasogastric feeding tubes in adults (interpretation of x ray images): summary of a safety report from the National Patient Safety Agency. BMJ. 2011 May 5;342:d2586. doi: 10.1136/bmj.d2586. No abstract available. PMID 21546422
- [Background] Parks J, Klaus S, Staggs V, Pena M. Outcomes of nasal bridling to secure enteral tubes in burn patients. Am J Crit Care. 2013 Mar;22(2):136-42. doi: 10.4037/ajcc2013105. PMID 23455863
- [Background] Puricelli MD, Newberry CI, Gov-Ari E. Avulsed Nasoenteric Bridle System Magnet as an Intranasal Foreign Body. Nutr Clin Pract. 2016 Feb;31(1):121-4. doi: 10.1177/0884533615611858. Epub 2015 Oct 20. PMID 26487513
- [Background] Seder CW, Janczyk R. The routine bridling of nasojejunal tubes is a safe and effective method of reducing dislodgement in the intensive care unit. Nutr Clin Pract. 2008 Dec-2009 Jan;23(6):651-4. doi: 10.1177/0884533608326139. PMID 19033225
- [Background] Seder CW, Stockdale W, Hale L, Janczyk RJ. Nasal bridling decreases feeding tube dislodgment and may increase caloric intake in the surgical intensive care unit: a randomized, controlled trial. Crit Care Med. 2010 Mar;38(3):797-801. doi: 10.1097/CCM.0b013e3181c311f8. PMID 19851098